CLINICAL TRIAL: NCT04466241
Title: Combination Therapies to Reduce the Nasopharyngeal Carriage of SARS-CoV-2 and Improve the Outcome of COVID-19 Infection in Ivory Coast (INTENSE-COV): a Phase IIb Randomized Clinical Trial
Brief Title: Combination Therapies to Reduce Carriage of SARS-Cov-2 and Improve Outcome of COVID-19 in Ivory Coast: a Phase Randomized IIb Trial
Acronym: INTENSE-COV
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: University of Bordeaux (Other); PACCI Program (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANRS COV01 INTENSE COV
Record Dates: First submitted 2020-07-06; First posted 2020-07-10 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: COVID-19; COVID-19 Drug Treatment; Severe Acute Respiratory Syndrome Coronavirus 2
Keywords: COVID-19; Combination therapy; Atorvastatin; Telmisartan; Lopinavir/ritonavir; SARS-COV-2; Viral load
MeSH Terms: conditions — COVID-19 | interventions — Lopinavir; Ritonavir; lopinavir-ritonavir drug combination; Telmisartan; Atorvastatin; Tablets

STUDY DESIGN:
Intervention Model Description: Phase IIb, comparative, multicenter, randomized, superiority, parallel-group, open-label clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Lopinavir/ritonavir (Active Comparator): Lopinavir boosted by ritonavir 200mg/50mg: 2 tablets morning and evening from Day 1 to Day 10
  Interventions: Drug: Lopinavir/Ritonavir 200 MG-50 MG Oral Tablet
- Lopinavir/ritonavir + telmisartan (Experimental): * Lopinavir boosted by ritonavir 200mg/50mg: 2 tablets morning and evening from Day 1 to Day 10
  * Telmisartan 40 mg : 1 tablet daily from Day 1 to Day 10
  Interventions: Drug: Lopinavir/Ritonavir 200 MG-50 MG Oral Tablet; Drug: Telmisartan 40Mg Oral Tablet
- Lopinavir/ritonavir + atorvastatin (Experimental): * Lopinavir boosted by ritonavir 200mg/50mg: 2 tablets morning and evening from Day 1 to Day 10
  * Atorvastatin 20 mg : 1 tablet daily from Day 1 to Day 10
  Interventions: Drug: Lopinavir/Ritonavir 200 MG-50 MG Oral Tablet; Drug: Atorvastatin 20 Mg Oral Tablet

INTERVENTIONS:
Drug: Lopinavir/Ritonavir 200 MG-50 MG Oral Tablet — 2 tablets morning and evening from Day 1 to Day 10
  Other Names: LPV/r; Aluvia
Drug: Telmisartan 40Mg Oral Tablet — 1 tablet daily from Day 1 to Day 10
  Other Names: TMS; Micardis; Pritor
  Arms: Lopinavir/ritonavir + telmisartan
Drug: Atorvastatin 20 Mg Oral Tablet — 1 tablet daily from Day 1 to Day 10
  Other Names: ATV; Tahor
  Arms: Lopinavir/ritonavir + atorvastatin

SUMMARY:
In January 2020, the new SARS-CoV-2 coronavirus was identified in China. The disease caused by this coronavirus was named COVID-19 by the World Health Organization (WHO). Since March 11, 2020, the WHO has described the global situation of COVID-19 as a pandemic. In Côte d'Ivoire, as in other African countries, the number of cases is increasing exponentially.

Coronaviruses are a family of viruses that cause illnesses ranging from the common cold to more severe pathologies. COVID-19 can result in fever or a feeling of fever (chills, hot-cold), cough, headache, aches and pains, unusual tiredness, sudden loss of smell, total disappearance of taste, or diarrhea. In severe forms, respiratory difficulties can lead to hospitalization in intensive care or even death.

Numerous studies are currently being conducted around the world to seek effective treatment, but few of them have started specifically in Africa. Moreover, most of these studies are using a single drug to control the infection, whether these are repositioned drugs, i.e. already being used for other diseases, or other newer drugs.

Currently in Côte d'Ivoire, the preferred treatment for COVID-19 is an antiviral: lopinavir/ritonavir (LPV/r), usually directed against the Human Immunodeficiency Virus (HIV).

Since the number of viruses (viral load) is high in the respiratory tract during COVID-19 infection, we propose in INTENSE-COV (ICOV) clinical trial to study whether the combination of two drugs is more effective than taking a single drug on reducing the viral load in the respiratory tract but also on reducing inflammation.

These drugs include the LPV/r already in use in Côte d'Ivoire as well as an antihypertensive drug - telmisartan, and a drug that lowers blood cholesterol - atorvastatin. All three have been known for a long time and have been shown to be effective against other viruses. In addition, they are generic, inexpensive and readily available in all countries.

The objectives of the ICOV study are therefore to improve viral eradication from the patient's body and respiratory tract, to reduce inflammation, to improve more rapidly the patient's state of health and to reduce the risk of transmission of the virus to others.

To participate in ICOV, patients must be over 18 years of age, have a COVID-19 infection confirmed by a specific test, have clinical manifestations of the infection, and have signed an informed consent. They will then be randomized into 3 treatment groups to ensure the robustness of the study results. The reference group will be treated with LPV/r, according to current recommendations in Côte d'Ivoire. The other 2 groups will be treated with LPV/r + telmisartan and LPV/r + atorvastatin respectively. The treatment will last 10 days and patients will be followed for a total of 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age.
* With SARS-CoV-2 infection confirmed by specific PCR.
* With clinical manifestations of the infection, such as fever or cough, or otolaryngologic (ORL) signs or respiratory difficulties, that started less than 7 days ago.
* COVID-19 specific treatment-naive.
* Women of childbearing age should accept the use of mechanical contraception during the study period.
* Informed consent signed by the patient.

Exclusion Criteria:

* Severe form of infection requiring oxygen therapy > 4l/min to achieve oxygen saturation > 94%.
* Patient whose weight is < 35kg.
* Pharmacological investigation contraindicating the introduction of a CYP450 inhibitor, in particular the CYP3A4 isoform.
* Known hypersensitivity to lopinavir, ritonavir, telmisartan, atorvastatin or their excipients.
* Renal impairment (eGFR <30 mL/min, CKD-EPI formulation).
* Known cirrhosis.
* Transaminases > 3N.
* Bilirubin > 2.6N.
* Electrocardiogram showing QTc> 500 ms.
* HIV-infected patient without treatment or treated with protease inhibitors (lopinavir, darunavir, atazanavir).
* Ongoing exposure to statins.
* Contraindications to the use of statin:

CPK > 5N, history of rhabdomyolysis or myopathies, increased risk when atorvastatin is administered with strong CYP3A4 inhibitors or transport proteins (cyclosporin, telithromycin, clarithromycin, delavirdine, stiripentol, ketoconazole, voriconazole, itraconazole, posaconazole, letermovir, erythromycin, diltiazem, verapamil, fluconazole).

* Ongoing exposure to sartans.
* Contraindications to the use of telmisartan:

patient on angiotensin-converting enzyme (ACE) inhibitors, aliskiren or other angiotensin receptor blockers (ARB).

* Curatorship or guardianship.
* Pregnancy or breastfeeding.
* Dementia or any other condition that prevents informed consent.
* Any reason that, at the discretion of the investigator, would compromise patient safety and cooperation in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Actual)
Dates: Start 2020-11-27 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with undetectable nasopharyngeal swab SARS-CoV-2 PCR and C-reactive protein (CRP) < 27 mg/L at Day 11 | Day 11

SECONDARY OUTCOMES:
Proportion of patients with clinical improvement on the 7-point ordinal scale at Day 11 and Day 28 | Day 11 and Day 28
Kinetics of SARS-CoV-2 viral load | Up to Day 28
Death rate at Day 11 and Day 28 | Day 11 and Day 28
All causes of death and Acute respiratory distress syndrome (ARDS) at Day 28 | Day 28
Time to hospital discharge | Up to Day 28
Duration of oxygen supplementation | Up to Day 28
Prevalence of grade III or IV adverse events | Up to Day 28
Residual concentration of lopinavir, telmisartan and atorvastatin | Up to Day 28
Evolution of inflammatory and immunological markers (CRP, fibrinogen, ferritin, d-dimer, dosing of IgG, IgA, IgM; TCD4, CD8, B lymphocytes, NK lymphocytes; naïve/memory T lymphocytes) | Up to Day 28
Evolution of endothelial activation markers (VEGF and soluble VEGF receptor,VE-cadherin, PECAM/CD31, CD42 and angiopoietin-2) | Up to Day 28
Proportion of patients with good results according to HIV status | Up to Day 28
Number of contact cases infected by COVID-19 at Day 28 | Day 28

CONTACTS AND LOCATIONS:
Locations (2):
- Côte d’Ivoire (2):
  - Service des Maladies Infectieuses et Tropicales, Centre Hospitalier et Universitaire (CHU) Treichville, Abidjan
  - Centre de Traitement des Maladies Infectieuses (CTMI), CHU de Yopougon, Abidjan

REFERENCES:
- [Background] Bonnet F, Doumbia A, Machault V, Ello FN, Bellecave P, Akpovo CB, Sidibe BT, Fernandez L, Kouame A, Adjogoua E, Dosso M, Niangoran S, Journot V, Eholie SP. Atorvastatin and telmisartan do not reduce nasopharyngeal carriage of SARS-CoV-2 in mild or moderate COVID-19 in a phase IIb randomized controlled trial. Sci Rep. 2024 Oct 23;14(1):25028. doi: 10.1038/s41598-024-72449-1. PMID 39443527